CLINICAL TRIAL: NCT04632797
Title: CROPSI Study A Randomized, Observer-blinded Clinical Trial Evaluating Effectiveness of Cryotherapy vs. Cryocompression for Preventing CIPN in Women Undergoing Chemotherapy
Brief Title: Cryotherapy vs. Cryocompression for Preventing Chemotherapy-induced-peripheral-neuropathy in Women Undergoing Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1224/2018
Record Dates: First submitted 2020-10-21; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Chemotherapeutic Toxicity; Chemotherapeutic Agent Toxicity
Keywords: Breast Cancer; Cervix Cancer; Endometrium Cancer; Ovarial Cancer; CIPN; Taxane
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: 1 to 1 randomization in either cryocompression or cryotherapy of the hands
Masking Description: It is an observer blinded study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryocompression (Active Comparator): Patients in this group receive cryocompression for the hands.
  Interventions: Device: Hilotherm Chemo Care
- Cryotherapy (Active Comparator): Patients in this group receive cryotherapy for the hands.
  Interventions: Device: Hilotherm Chemo Care

INTERVENTIONS:
Device: Hilotherm Chemo Care — Application of Hilotherm Chemo Care gloves for constant cryotherapy during chemotherapy application.

SUMMARY:
This study's aim is to show a benefit of Cryocompression (cooling hands with additional compression of the hands) in comparison to Cryotherapy (just cooling hands) in female cancer patients (with gynecological cancer) receiving chemotherapy with taxanes.

Patients who are not eligible for either cryocompression or cryotherapy are included in a control group.

The expected benefits with additional compression to the cryotherapy are reduction of chemotherapy induced polyneuropathy and reduced nail changes.

DETAILED DESCRIPTION:
In this randomized, observer blinded, monocentric study 196 patients will be included in a four years period.

The patients will be 1 to 1 randomized in either cryocompression or cryotherapy. Patients who are not eligible for either cryocompression or cryotherapy will be included in the control group.

Additionally every patient (excluding the control group) receives cryotherapy for the feet.

Before receiving the first chemotherapy CTCAE, Semmes-Weinstein monofilament examination (SWME), vibration test for hand and feet, and nerve conduction velocity (NCV) only for hands.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer or other gynecological tumors
* planned neoadjuvant, adjuvant or palliative chemotherapy
* </= two lines chemotherapy as pre-therapy (adjuvant chemotherapy counts as one line)
* at least three cycles of chemotherapy with taxanes
* written consent
* 18 years and older

Exclusion Criteria:

* PNP >/= 2
* neuralgia
* metastases in bones, metastases in soft tissue (located in skin, hands or feet)
* Raynaud syndrome
* peripheral arterial ischemia
* hand-feet syndrome

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-02-03 (Estimated); Study Completion 2024-02-03 (Estimated)

PRIMARY OUTCOMES:
NCV (nerve conduction velocity) | 4 years
  Comparison of efficacy of cryotherapy vs. cryocompression regarding occurence of ≥ CIPN III°
CTCAE 4.03 | 4 years
  Comparison of efficacy of cryotherapy vs. cryocompression regarding occurence of ≥ CIPN III°
SWME (Semmes Weinstein monofilament examination) | 4 years
  Comparison of efficacy of cryotherapy vs. cryocompression regarding occurence of ≥ CIPN III°
tuning-fork-test | 4 years
  Comparison of efficacy of cryotherapy vs. cryocompression regarding occurence of ≥ CIPN III°
EORTC QoLCIPN20 | 4 years
  Patient-reported outcomes (PRO)
Neuro-QoL Domain for Upper Extremity (FineMotor, ADL) | 4 years
  Patient-reported outcomes (PRO)

SECONDARY OUTCOMES:
National Cancer Institute Common Toxicity Criteria version 2 | 4 years
  Changes of nails
time frame until polyneuopathy occurs | 4 years
  time frame until polyneuopathy occurs whilst receiving Taxanes

CONTACTS AND LOCATIONS:
Overall Officials: Christine Brunner, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: Undecided